CLINICAL TRIAL: NCT01730703
Title: Why Join a Walking Program?
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 815599
Record Dates: First submitted 2012-11-09; First posted 2012-11-21 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Older Adults
Keywords: walking; incentives; elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults ages 65 and older

SUMMARY:
The purpose of this interview study is to learn why adults would join a walking program. This study involves interviews with persons who are 65 years of age or older. The interview takes approximately 25 minutes. A total of 132 people will be enrolled. This study will examine the utility or value of various potential features of an incentive-based walking program. These data will enable us to monitor and improve upon enrollment of incentive-based walking programs.

ELIGIBILITY:
Inclusion Criteria:

* age 65 or older
* self rated health at least good on a scale of poor, fair, good, very good, excellent
* self reports no physical reason not to exercise or health condition that would interfere with being active
* self reports able to walk at least 2 blocks without assistance or stopping not participating in a daily walking exercise program

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Adults ages 65 and older who are generally in good health and are not enrolled in daily walking exercise programs, and are able to provide their own verbal informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Willingness to Participate | Participation in the study will include only one interview, lasting approximately 25 minutes. Willingness to participate will be assessed during this first and only interview with the participant.
  The goal of this pilot project is to examine why adults would join an incentive-based walking program. Our focus is willingness to participate. Willingness to participate is measured on a 7 point ordinal scale.

SECONDARY OUTCOMES:
Self explicated conjoint task | Participation in the study will include only one interview, lasting approximately 25 minutes. The self explicated conjoint task will be assessed during this first and only interview with the participant.
  This study will examine the utility or value of various potential features of an incentive-based walking program. These data will enable us to monitor and improve upon enrollment of incentive-based walking programs.
  How important is this feature? How desirable is this feature?
  Importance: 7 point ordered scale from "extremely" to "not at all" Desirability: 7 point from "very desirable" to "very undesirable"

CONTACTS AND LOCATIONS:
Overall Officials: Jason Karlawish, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States